CLINICAL TRIAL: NCT07153367
Title: Using a Fixed Dosage of Follitropin Delta for Ovarian Stimulation for Intrauterine Insemination: Rekovelle for Intrauterine Successful Experience (RISE)
Acronym: RISE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RISE
Record Dates: First submitted 2025-07-03; First posted 2025-09-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Infertility; Insemination
MeSH Terms: conditions — Infertility | interventions — follitropin delta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rekovelle Arm (Experimental)
  Interventions: Drug: REKOVELLE (Follitropin Delta)

INTERVENTIONS:
Drug: REKOVELLE (Follitropin Delta) — Each patient will start the ovarian stimulation with a fixed dose of 3,66 mcg of Rekovelle ® on day 4 of the natural cycle (Stimulation day 1-S1). The stimulation period will last a maximum of 13 days.
  Patients will be regularly evaluated to monitor the response to stimulation with ultrasound scan and blood sampling

SUMMARY:
The aim of this study is to evaluate the use of a fixed dose of 3.66 mcg of follitropin delta (Rekovelle) on ovarian response during ovarian stimulation for intrauterine insemination (IUI). The assumption is that this fixed dose will be effective while minimizing the risk of multiple pregnancies. A recent study demonstrated the efficacy of follitropin delta for ovarian stimulation in IUI, and it has been approved in France for controlled ovarian stimulation in assisted reproductive techniques such as in vitro fertilization (IVF) and IVF with intracytoplasmic sperm injection (ICSI). With an adapted dose of Rekovelle for patients with regular menstrual cycles, ovarian stimulation is optimized from the first attempt, promoting the development of two follicles to improve pregnancy chances while reducing the risk of multiple pregnancies. This approach aims to achieve pregnancy faster and provide a more comfortable treatment experience.

DETAILED DESCRIPTION:
Intrauterine insemination (IUI) is a frequently used step in the management of unexplained infertility or mild fertility disorders. In normal-weight patients, the main objective of ovarian stimulation in IUI is to obtain a controlled ovarian response, ideally bifollicular.

Moreover, the main risks currently associated with IUI are multiple pregnancies and iatrogenic complications (cycle cancellation due to insufficient response or excessive response to stimulation more than 3 follicles). It is therefore essential to optimize stimulation treatment protocols to ensure IUI under the best possible conditions.

Due to a precise dose adjustment with Follitropin Delta, the product used in the study (REKOVELLE), for normo-ovulatory patient, an optimal response (bifollicular response) is expected for the majority of patients from the first stimulation. This goal will also facilitate quicker pregnancy attainment and reduce the risk of drop-out and insémination annulation The hypothesis is that this dosage would be efficient and also minimize the risk of multiple pregnancies During the screening visit, the investigator checks the patient's eligibility and informs her about the RISE study. At the inclusion visit, written informed consent is obtained, and the Rekovelle® treatment is explained and initiated. Monitoring visits start on day 9 and then every 2 days until two mature follicles develop. Ovocyte maturation is triggered with an hCG injection, followed by insemination 36 hours later, performed according to routine care. Follow-up visits occur at 6-8 weeks and 13 weeks post-insemination.

ELIGIBILITY:
Inclusion Criteria:

* Normo-ovulatory patients
* 18 - 38 included years old
* BMI between 18 and 29 included kg/m²
* Regular menstrual cycles
* At least one healthy Fallopian tube
* Normal uterus cavity
* First treatment for IUI
* Affiliation to the social security

Exclusion Criteria:

* Endometriosis Stage III
* Total mobile sperm count <1 million
* Severe spermatogenesis disorders
* Women with Poly Cystic Ovary Syndrom
* History of OHSS or excessive response to gonadotrophins
* Chronic disease with contraindication to ovarian stimulation with gonadotrophins
* Known genetic disease
* Hypothalamus or pituitary tumors
* Ovarian hypertrophy or ovarian cyst not due to polycystic ovary syndrome
* Gynecological bleeding of unknown etiology
* Ovarian, uterine or breast carcinoma
* Primary ovarian failure
* Genital malformations incompatible with pregnancy
* Uterine fibroids incompatible with pregnancy
* Protected persons (pregnant women, nursing mothers, person under guardianship, minors, persons deprived of liberty, and persons unable to give consent)
* Tumors (including meningioma) whose development is known or suspected to be progesterone-dependent
* History of hepatic dysfunction
* Have been receiving progestogen therapy for more than 6 months
* Known contraindication to hormonal treatments (progestogens or oestrogens), or with a history of adverse events related to their use
* Previous thromboembolism events during or following the use of gonadotrophins or with high risk factors for thromboembolic events (venous or arterial)
* Hypersensitivity to the active substance or to any of the excipients
* High risk of OHSS such as women with AMH ≥ 35 pmol/L
* History of severe uterine malformation (unicornuate or bicornuate uterus),
* Past history of ovarian torsion
* Uncontrolled thyroid dysfunction
* Uncontrolled adrenal dysfunction
* Hydrosalpynx
* Breast pathologies not compatible with gonadotrophin stimulation
* Use of infertility medications that could affect follicle stimulation and maturation such as GH
* Participation in other interventional research
* Not able to understand and sign the written informed consent form

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Des femmes
Enrollment: 80 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2027-12-17 (Estimated); Study Completion 2028-03-17 (Estimated)

PRIMARY OUTCOMES:
Percentage of cycles with two mature follicles (total of two ovaries) at the stage of triggering ovulation | up to 9 months
  Percentage of cycles with two mature follicles (total of two ovaries) at the stage of triggering ovulation (follicles diameter ≥14 mm) and no follicles between 10 et 13 mm.

SECONDARY OUTCOMES:
Number of follicles ≥14 mm on the day of trigger | Up to Day 15 of the cycle (each cycle is 28 days)
  Number of follicles ≥14 mm on the day of trigger ( by cycle)
Number of follicles between 10 et 13 mm on the day of trigger | Up to Day 15 of the cycle (each cycle is 28 days)
  Number of follicles between 10 et 13 mm on the day of trigger (by cycle)
Percentage of cycles with two mature follicles (total of two ovaries) at the stage of triggering ovulation (follicles diameter ≥14 mm) and no follicles between 10 et 13 mm for each cycle and according to dose adjustment | up to 9 months
  Percentage of cycles with two mature follicles (total of two ovaries) at the stage of triggering ovulation (follicles diameter ≥14 mm) and no follicles between 10 et 13 mm for each cycle and according to dose adjustment
Presence or absence of dose adjustment in subsequent cycles | up to 9 months
  Presence or absence of dose adjustment in subsequent cycles
E2 level on the day of trigger | Up to Day 15 of the cycle (each cycle is 28 days)
  E2 level on the day of trigger (pg/ml)
Dose adjustment on subsequent cycle(s) : quantity of mcg | up to 9 months
  Dose adjustment on subsequent cycle(s) : quantity of mcg
PG level on the day of trigger | Up to Day 15 of the cycle (each cycle is 28 days)
  PG level on the day of trigger (ng/ml)
LH level on the day of trigger | Up to Day 15 of the cycle (each cycle is 28 days)
  LH level on the day of trigger (UI/L)
Frequency of spontaneous LH surge by cycle , at the end of stimulation | up to 9 months
  Frequency of spontaneous LH surge by cycle , at the end of stimulation (last day of stimulation)
Cycle cancellation rate | up to 9 months
  Cycle cancellation rate (by cycle) . The Cycle is cancelled when more than 2 follicles ≥ 14mm or 4 follicles ≥ 10mm, or if there is no response to treatment.
Pregnancy loss rate | up to 9 months
  Pregnancy loss rate
Rate of Biochemical pregnancy (βhCG test) by initiated cycle | From enrollment to 2 weeks after IUI
  Rate of Biochemical pregnancy (βhCG test) by initiated cycle
Rate of Clinical pregnancy by initiated cycle | From enrollment to 8 weeks after IUI
  Rate of Clinical pregnancy by initiated cycle
Rate of Ongoing pregnancy by initiated cycle | From enrollment to 13 weeks after IUI
  Rate of Ongoing pregnancy by initiated cycle
Pregnancy rate with one follicle or two follicles diameter ≥14 mm | up to 9 months
  Pregnancy rate with one follicle or two follicles diameter ≥14 mm
Multiple pregnancy rate | up to 9 months
  Multiple pregnancy rate
Time to pregnancy | From first stimulation until pregnancy confirmed by HCG > 100 UI/L, assessed up to 6 months.
  Time to pregnancy (time between 1st stimulation and date of pregnancy)
The number of stimulation days. | up to 9 months
  The number of stimulation days.
Unexpected and related Events | up to 9 months
  Unexpected and related Events
Duration in days between each cycle | up to 9 months
  Duration in days between each cycle
Dose adjustment on subsequent cycle(s) : number of cycles | up to 9 months
  Dose adjustment on subsequent cycle(s) : number of cycles
Dose adjustment on subsequent cycle(s) : percentage of cycles | up to 9 months
  Dose adjustment on subsequent cycle(s) : percentage of cycles
Rate of Biochemical pregnancy (βhCG test) by insemination | From enrollment to 2 weeks after IUI
  Rate of Biochemical pregnancy (βhCG test) by insemination
Rate of Biochemical pregnancy (βhCG test):cumulative rates | From enrollment to 2 weeks after IUI
  Rate of Biochemical pregnancy (βhCG test) : cumulative rates
Rate of Clinical pregnancy by insemination | From enrollment to 8 weeks after IUI
  Rate of Clinical pregnancy by insemination
Rate of Clinical pregnancy (cumulative rates) | From enrollment to 8 weeks after IUI
  Rate of Clinical pregnancy (cumulative rates)
Rate of Ongoing pregnancy by insemination | From enrollment to 13 weeks after IUI
  Rate of Ongoing pregnancy by insemination
Rate of Ongoing pregnancy: cumulative rates | From enrollment to 13 weeks after IUI
  Rate of Ongoing pregnancy: cumulative rates
The duration of stimulation for each cycle | up to 9 months
  The duration of stimulation for each cycle
Endometrial thickness | up to 9 months
  Endometrial thickness
Pregnancy outcome according to the cycle rank | up to 9 months
  Pregnancy outcome according to the cycle rank
Cumulative pregnancy outcome up to 3 cycles | up to 9 months
  Cumulative pregnancy outcome up to 3 cycles
Number of OHSS | up to 9 months
  Number of OHSS
Number of ectopic pregnancy | up tp 9 months
  Number of ectopic pregnancy
Number of ovarian torsion | up to 9 months
  Number of ovarian torsion
Number of thromboembolic events | up to 9 months
  Number of thromboembolic events
Causes of cycle cancellation | up to 9 months
  Causes of cycle cancellation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Chevalier, Principal Investigator — Centre AMP Saint Roch
Locations (5):
- France (5):
  - Cabinet Dr Elodie Descat-Polyclinique Jean Villar, Bruges
  - Chi Creteil, Créteil
  - Cabinet Dr Géraldine PORCU-Institut de Médecine de la Reproduction, Marseille
  - Cabinet Dr Nicolas Chevalier-Centre AMP Saint Roch, Montpellier
  - Cabinet Dr Nathalie Massin- Hôpital Américain De Paris, Neuilly-sur-Seine

IPD SHARING:
Plan to Share IPD: No